CLINICAL TRIAL: NCT03595644
Title: Maintenance Targeted Therapy With or Without Stereotactic Body Radiation Therapy for Stage IV Non-small Cell Lung Cancer: a Prospective, Multicenter, Randomized Controlled Clinical Trial.
Brief Title: Maintenance Targeted Therapy With or Without Stereotactic Body Radiation Therapy for Stage IV Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tongji Hospital (Other)
Collaborators: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Renmin Hospital of Wuhan University (Other); Wuhan University (Other); Hubei Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TJCC-LC001
Record Dates: First submitted 2018-06-19; First posted 2018-07-23 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Stage IV Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SBRT plus TKI group (Experimental): SBRT with photon and dose is 40-50Gy/5F after three months after EGFR-TKI treatment
  Interventions: Radiation: SBRT+TKI
- TKI treatment group (Active Comparator): Standard EGFR-TKI(Gefitinib, erlotinib or icotinib) Gefitinib: 250mg po Qd Erlotinib: 150mg po Qd Icotinib: 125mg po tid
  Interventions: Drug: TKI

INTERVENTIONS:
Radiation: SBRT+TKI — Received SBRT after three months after EGFR-TKI treatment
  Arms: SBRT plus TKI group
Drug: TKI — Received EGFR-TKI treatment
  Arms: TKI treatment group

SUMMARY:
This is a Prospective, Multicenter, Randomized Controlled study to evaluate Stereotactic Body Radiation Therapy (SBRT) as a potential treatment for stage IV non-small cell lung cancer (NSCLC) that has a mutated epidermal growth factor receptor (EGFR) and has been receiving treatment with a targeted agent such as gefitinib, erlotinib and icotinib.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have biopsy proven metastatic NSCLC (Stage IV).
2. Patients must have received first line chemotherapy, from 4-6 cycles, and achieved stable disease or a partial response.
3. Patients receiving first-line erlotinib, gefitinib, or icotinib for EGFR mutant-positive for 3 months and achieved stable disease, partial response or completely response.
4. Age 18 to 75 years old.
5. Patients must have measurable disease at baseline.
6. The amount of metastatic focus <5.
7. ECOG score 0-2
8. Adequate normal organ and marrow function for TKI treatment and radiotherapy.
9. Patients must has sensitizing EGFR mutation (e.g. exon 19 deletion or exon 21 L858R)
10. Patients must provide written informed consent to participate in the study.

Exclusion Criteria:

1. Patients who previously received radiotherapy to the primary site.
2. Patient can't tolerate radiotherapy or targeted therapy;
3. Pregnant or nursing women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2017-02-12 (Actual); Primary Completion 2019-06-10 (Actual); Study Completion 2020-12-10 (Actual)

PRIMARY OUTCOMES:
PFS | 2 years
  Progression-free survival: From the first treatment to the date of first documentation of disease progression, or death due to any cause

SECONDARY OUTCOMES:
OS | 3 year
  Overall survival: From the first administration to death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: li Zhang, MD,PhD, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital of Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Iyengar P, Wardak Z, Gerber DE, Tumati V, Ahn C, Hughes RS, Dowell JE, Cheedella N, Nedzi L, Westover KD, Pulipparacharuvil S, Choy H, Timmerman RD. Consolidative Radiotherapy for Limited Metastatic Non-Small-Cell Lung Cancer: A Phase 2 Randomized Clinical Trial. JAMA Oncol. 2018 Jan 11;4(1):e173501. doi: 10.1001/jamaoncol.2017.3501. Epub 2018 Jan 11. PMID 28973074
- [Background] Gomez DR, Blumenschein GR Jr, Lee JJ, Hernandez M, Ye R, Camidge DR, Doebele RC, Skoulidis F, Gaspar LE, Gibbons DL, Karam JA, Kavanagh BD, Tang C, Komaki R, Louie AV, Palma DA, Tsao AS, Sepesi B, William WN, Zhang J, Shi Q, Wang XS, Swisher SG, Heymach JV. Local consolidative therapy versus maintenance therapy or observation for patients with oligometastatic non-small-cell lung cancer without progression after first-line systemic therapy: a multicentre, randomised, controlled, phase 2 study. Lancet Oncol. 2016 Dec;17(12):1672-1682. doi: 10.1016/S1470-2045(16)30532-0. Epub 2016 Oct 24. PMID 27789196
- [Background] de Vin T, Engels B, Gevaert T, Storme G, De Ridder M. Stereotactic radiotherapy for oligometastatic cancer: a prognostic model for survival. Ann Oncol. 2014 Feb;25(2):467-71. doi: 10.1093/annonc/mdt537. Epub 2013 Dec 18. PMID 24355488
- [Derived] Peng P, Gong J, Zhang Y, Zhou S, Li Y, Han G, Meng R, Chen Y, Yang M, Shen Q, Chu Q, Xia S, Zhang P, Zhang L, Chen Y, Zhang L. EGFR-TKIs plus stereotactic body radiation therapy (SBRT) for stage IV Non-small cell lung cancer (NSCLC): A prospective, multicenter, randomized, controlled phase II study. Radiother Oncol. 2023 Jul;184:109681. doi: 10.1016/j.radonc.2023.109681. Epub 2023 Apr 25. PMID 37105304